CLINICAL TRIAL: NCT07167693
Title: Phase 1 Randomized Clinical Trial of Arginine Hydrochloride Administration to Reduce Duration of Diabetic Ketoacidosis in Patients With Type 2 Diabetes
Brief Title: Phase 1 Trial of Arginine Hydrochloride for the Management of Diabetic Ketoacidosis in Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David K Carroll (Other)
Collaborators: Wayne State University (Other); Detroit Medical Center (Other)
Responsible Party: Sponsor-Investigator, David K Carroll, Assistant Professor of Emergency Medicine, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-12-7395
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes (DM); Diabetic Ketoacidosis; Ketosis Prone Diabetes; Hyperglycaemia (Diabetic)
Keywords: Arginine hydrochloride; Arginine; R-Gene 10; Insulin secretagogue; Endogenous insulin secretion; C-peptide; C-peptide to glucose ratio; Type 2 ketosis-prone diabetes (T2KPD); Flatbush diabetes; Ketosis-prone diabetes (KPD); Hyperglycemic crisis; Nitric oxide (NO); Global arginine bioavailability ratio (GABR); Mitochondrial function
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Ketoacidosis; Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Arginine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel two-arm assignment in the emergency department. Each participant receives a single, 30-minute IV infusion as early as feasible after DKA is recognized, in addition to standard DKA care directed by the treating team. Arms: (1) arginine hydrochloride 30 g in 300 mL (R-Gene® 10) and (2) matching placebo (0.9% saline). No clinical care elements are withheld or mandated. Primary biomarker time points occur 10, 30 (end of infusion), and 90 minutes from infusion start; secondary outcomes include β-hydroxybutyrate clearance and total insulin dose in the first 24 h. Adults with suspected/confirmed ketosis-prone type 2 DKA are enrolled across four Detroit-area hospitals.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple-blind with centralized 1:1 allocation concealment. A site research pharmacist (unblinded) prepares study drug; infusion containers are covered to mask volume/appearance and both arms are run over 30 minutes using identical pump settings. Participants, bedside clinicians, investigators, and outcomes assessors remain blinded through database lock. Emergency unblinding is permitted for medical necessity via pharmacy access to allocation codes; all unblindings are logged. Laboratory personnel analyze specimens using coded IDs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arginine Hydrochloride 30 g IV + Standard DKA Care (Active Comparator): Single, blinded 30-minute intravenous infusion of arginine hydrochloride 30 g/300 mL (R-Gene® 10), initiated as early as feasible after recognition of DKA, in addition to standard DKA management (fluids, insulin, electrolytes) at the treating clinician's discretion. Infusion procedures are matched to placebo (covered containers; standardized pump settings) to maintain blinding. Study blood draws occur at 0 (pre-infusion), 10, 30, and 90 minutes for C-peptide/glucose and targeted amino acids; clinical labs are used to assess β-hydroxybutyrate clearance and total insulin administered in the first 24 h.
  Interventions: Drug: Arginine hydrochloride
- Placebo (0.9% Saline) IV + Standard DKA Care (Placebo Comparator): Single, blinded 30-minute intravenous infusion of matching placebo: 0.9% sodium chloride (normal saline) in a 500 mL container, administered at a standardized rate to mimic the active arm, plus standard DKA management directed by the treating team. Appearance and administration procedures match the arginine arm (covered containers; identical pumps/tubing) to preserve blinding. Study blood draws and assessments occur on the same schedule as the arginine arm (0, 10, 30, and 90 minutes).
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Arginine hydrochloride — Single intravenous infusion of arginine hydrochloride 30 g in 300 mL 10% solution (R-Gene® 10), administered over 30 minutes via infusion pump. Given as early as feasible after recognition of DKA and in addition to standard DKA care (fluids, insulin, electrolytes) at the treating clinician's discretion. Investigational pharmacy prepares and dispenses blinded study drug; containers are covered to mask appearance and infusion parameters match placebo. Continuous safety monitoring with prespecified stop criteria. Study blood draws at 0 (pre-infusion), 10, 30, and 90 minutes for C-peptide/glucose and amino acids; clinical labs track β-hydroxybutyrate clearance and total insulin over 24 hours.
  Other Names: L-arginine hydrochloride; Arginine HCl; R-Gene 10; Arginine hydrochloride injection 10%
  Arms: Arginine Hydrochloride 30 g IV + Standard DKA Care
Drug: Sodium Chloride 0.9% — Placebo comparator: 0.9% sodium chloride administered as a single 30-minute intravenous infusion using identical tubing, pump settings, and covered container as the active arm to preserve blinding. Initiated as early as feasible after recognition of DKA and provided in addition to standard DKA care at the treating clinician's discretion. Study assessments occur on the same schedule as the active arm (0, 10, 30, and 90 minutes) with continuous safety monitoring during and after infusion and follow-up through 90 days.
  Other Names: Normal saline
  Arms: Placebo (0.9% Saline) IV + Standard DKA Care

SUMMARY:
Diabetic ketoacidosis (DKA) is increasingly recognized in adults with "ketone-prone" type 2 diabetes. In many of these patients, the pancreas can still make insulin but becomes temporarily "stunned" during severe, prolonged high blood sugar. Arginine is a naturally occurring amino acid that can trigger the pancreas to release its own insulin when glucose is high. It is FDA-approved for other uses and has been given intravenously for decades with a strong safety record. Whether a single arginine infusion given early during DKA can safely boost the body's insulin and speed recovery has not been tested.

This randomized, double-blind, placebo-controlled, phase 1/2 trial will enroll 60 adults who present to one of four Detroit-area emergency departments with DKA consistent with ketone-prone type 2 diabetes (high glucose and significant ketones). Participants will receive standard DKA care ordered by their clinicians. In addition, under blinded conditions they will receive either arginine hydrochloride 30 grams (in 300 mL) or placebo (normal saline), infused intravenously over 30 minutes as early as feasible after DKA is recognized.

The main question is whether arginine increases endogenous (self-made) insulin soon after infusion. We will measure C-peptide (a marker released in equal amounts with insulin) and glucose at 10, 30, and 90 minutes after the start of the infusion and calculate the C-peptide/glucose ratio. Secondary measures include the rate of ketone (β-hydroxybutyrate) clearance and the total insulin dose required in the first 24 hours. Additional blood tests will examine arginine and related amino acids, and a small sample of platelets will be used to explore mitochondrial function. Safety will be closely monitored during and after the infusion, and participants will be contacted at 90 days to assess for any delayed problems.

Potential risks include temporary flushing, nausea, or headache; the infusion can be stopped at any time if needed. Potential benefits include faster resolution of ketosis and reduced insulin needs, but benefits cannot be guaranteed for individual participants.

DETAILED DESCRIPTION:
Background and Rationale. A substantial subset of adults with type 2 diabetes develop DKA ("ketone-prone" type 2 diabetes). Many of these patients lack diabetes autoantibodies (A-) and retain recoverable β-cell function (β+). The pathophysiology appears to involve reversible β-cell dysfunction from prolonged hyperglycemia. Arginine, a cationic amino acid and physiologic insulin secretagogue, depolarizes β-cells and enhances glucose-dependent insulin release within minutes. Prior human studies show prompt rises in insulin and C-peptide after arginine in individuals with preserved β-cell reserve. Arginine may also improve nitric-oxide bioavailability and mitigate mitochondrial dysfunction-processes implicated in hyperglycemic crises. We therefore hypothesize that early intravenous arginine, added to usual DKA care, will acutely increase endogenous insulin secretion and speed clearance of ketosis without added safety concerns.

Design and Setting. Prospective, phase 1/2, randomized, double-blind, placebo-controlled, parallel-group trial at four emergency departments in the Detroit metropolitan area. Target enrollment is 60 participants (1:1 allocation).

Participants. Adults (>17 years) with hyperglycemia (generally ≥250 mg/dL) and significant ketonemia/ketosis consistent with DKA and a clinical phenotype of ketone-prone type 2 diabetes. Key exclusions include known type 1 diabetes or positive GAD65 antibodies, chronic dialysis, cirrhosis, pregnancy, allergy to arginine, or features of moderate/greater alcohol intoxication. Screening may use point-of-care capillary β-hydroxybutyrate (BHB) or breath acetone to expedite identification; confirmatory laboratory thresholds will be used per protocol.

Intervention. As early as logistics allow after recognition of DKA, participants will receive a blinded 30-minute intravenous infusion of either arginine hydrochloride 30 g in 300 mL (R-Gene® 10) or matching placebo (normal saline 500 mL). Treating teams will manage DKA per standard institutional protocols; the study does not restrict clinical care (fluids, insulin, electrolytes).

Outcomes.

Primary endpoint: Endogenous insulin secretion quantified by the C-peptide/glucose ratio at 10, 30 (end of infusion), and 90 minutes after infusion start.

Key secondary endpoints: (a) Rate of BHB decline (ketone clearance), and (b) total insulin administered in the first 24 hours.

Mechanistic/biomarker endpoints: Plasma amino acids-especially arginine, citrulline, and ornithine-to compute the Global Arginine Bioavailability Ratio (arginine/[ornithine+citrulline]) at baseline and 90 minutes; insulin, proinsulin, and diabetes autoantibodies. Exploratory endpoint: Platelet mitochondrial complex IV and V activities as markers of oxidative phosphorylation.

Safety Monitoring. Participants will be observed closely during and after infusion with serial vital signs and symptom checks (e.g., flushing, nausea, headache). Pre-specified stop criteria allow immediate interruption of the infusion. Adverse events will be assessed to 90 days (telephone/medical record review) and reported per regulatory guidance. Because of the small size and favorable safety profile of intravenous arginine, the study qualifies as early-phase with streamlined oversight; an independent Data and Safety Monitoring Board has nonetheless been chartered.

Sample Size and Analysis. Based on prior insulinotropic responses to arginine, we powered the study to detect a moderate-to-large effect (standardized mean difference ~0.8) in the primary endpoint with 80% power and α=0.05, yielding ~26 per group. Allowing for attrition, we plan to enroll 60 participants. The C-peptide/glucose ratio will be assessed for normality and compared between groups with appropriate parametric or transformed analyses; ketone clearance and insulin dose will be analyzed similarly. Prespecified sensitivity analyses will account for baseline severity and timing of insulin initiation.

Operational Notes. To facilitate early enrollment, research staff will screen patients with suspected DKA using point-of-care BHB or breath acetone while confirmatory labs are pending. Blood draws for study assays occur at baseline (pre-infusion), 10, 30, and 90 minutes, with additional clinically obtained labs used for outcomes (e.g., BHB over the first 24 hours). Platelet-rich plasma will be stored for exploratory mitochondrial testing using validated methods.

Impact. If early arginine infusion safely augments endogenous insulin and accelerates ketone clearance, this pragmatic, low-cost, readily available therapy could reduce reliance on prolonged insulin infusions, shorten ICU/ED resource use, and improve patient experience during DKA. Findings will inform the design of a larger phase 2/3 trial focused on clinical effectiveness and health-system outcomes in ketone-prone type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years.
* Unscheduled presentation to a participating emergency department with hyperglycemia (serum glucose >250 mg/dL) and significant ketonemia consistent with DKA, defined as laboratory serum/plasma β-hydroxybutyrate (BHB) >20 mg/dL (≈≥1.9 mmol/L).

Note: point-of-care capillary BHB ≥1.5 mmol/L and/or breath acetone ≥0.01% may be used for screening while confirmatory labs are pending; if confirmatory BHB ≤20 mg/dL, the participant is a screen failure.

* Clinical phenotype consistent with ketosis-prone type 2 diabetes (no known prior diagnosis of type 1 diabetes).
* Able to provide written informed consent and comply with study procedures in the ED.

Exclusion Criteria:

* Current renal replacement therapy for chronic kidney disease (hemodialysis or peritoneal dialysis).
* Known history of type 1 diabetes mellitus or known GAD65 autoantibody positivity.
* Diagnosed cirrhosis/advanced chronic liver disease.
* Pregnancy (known pregnancy or positive test at screening).
* Known allergy or hypersensitivity to arginine or its components.
* Features of at least moderate acute alcohol intoxication at screening, per treating team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in endogenous insulin secretion (C-peptide/glucose ratio) | Baseline (pre-infusion) to 90 minutes after infusion start
  Serum C-peptide (ng/mL) and plasma glucose (mg/dL) will be measured at 0 (pre-infusion), 10, 30, and 90 minutes from infusion start. The C-peptide/glucose ratio will be calculated at each time. Primary summary = change from baseline to 90 minutes (90-min ratio minus baseline ratio). Higher values indicate greater recruitable endogenous insulin secretion.

SECONDARY OUTCOMES:
Change in beta-hydroxybutyrate (BHB) concentration | Baseline to 24 hours
  Difference in serum BHB from baseline to 24 hours (baseline BHB minus 24-hour BHB). Positive values reflect ketone clearance.
Rate of BHB clearance | 0-24 hours
  Slope of BHB concentration over time using all clinically obtained values in the first 24 hours.
Total insulin administered in first 24 hours | 0-24 hours
  Sum of all insulin doses (IV and/or subcutaneous) administered as part of routine care.
Plasma arginine concentration (change from baseline) | Baseline to 90 minutes
  HPLC-based quantification of plasma arginine at baseline and 90 minutes; change = 90-min minus baseline.
Global Arginine Bioavailability Ratio (GABR) | Baseline to 90 minutes
  GABR = [arginine]/([ornithine]+[citrulline]); change from baseline to 90 minutes.

OTHER OUTCOMES:
Platelet mitochondrial complex IV activity (change from baseline) | Baseline to 90 minutes
  Enzymatic activity of cytochrome c oxidase (complex IV) measured in isolated platelet-rich plasma; normalized to protein content or citrate synthase as per lab SOP; change = 90-min minus baseline.
Platelet mitochondrial complex V (ATP synthase) activity (change from baseline) | Baseline to 90 minutes
  Activity measured in isolated platelets; normalized per lab SOP; change = 90-min minus baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the primary and secondary outcomes, including: demographics (age, sex), baseline clinical values, all C-peptide and glucose measurements at 0/10/30/90 minutes, β-hydroxybutyrate values used to derive ketone-clearance metrics, total insulin administered in the first 24 hours, adverse events, and (when available) amino-acid measures and platelet mitochondrial assays. A data dictionary will accompany the dataset. All IPD will be de-identified consistent with HIPAA Safe Harbor (direct identifiers removed; dates converted to study day/time; site identifiers suppressed).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning after publication of the primary results manuscript (or within 24 months of last-patient last-visit, whichever occurs first) and available for at least 5 years thereafter.
Access Criteria: Access is provided upon reasonable request to the Study Contact listed on this record. Requestors must submit a brief proposal with analysis aims and statistical plan and provide evidence of IRB/ethics review or exemption. A Data Use Agreement is required (no re-identification, no onward sharing, secure storage, and acknowledgment of the source in resulting works). Approved requests will receive the de-identified dataset and data dictionary via secure transfer. Aggregated results will also be made available on reasonable request.